CLINICAL TRIAL: NCT04261855
Title: A Phase Ib/II Study of Combination Avelumab With Peptide Receptor Radionuclide Therapy or Conventional Fractionated Radiotherapy in Patients With Metastatic Merkel Cell Carcinoma
Brief Title: Targeted Therapy and Avelumab in Merkel Cell Carcinoma
Acronym: GoTHAM
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Melanoma and Skin Cancer Trials Limited (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10.17
Record Dates: First submitted 2020-02-06; First posted 2020-02-10 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Metastatic Merkel Cell Carcinoma
Keywords: radiotherapy; peptide receptor radionuclide therapy; neuroendocrine tumour; rare cancer; merkel cell; carcinoma; immunotherapy; merkel cell carcinoma
MeSH Terms: conditions — Carcinoma, Merkel Cell; Neuroendocrine Tumors; Carcinoma | interventions — avelumab; Radiotherapy; Lutetium-177; lutetium Lu 177 dotatate

STUDY DESIGN:
Intervention Model Description: The LuTate treatment arm is now closed to recruitment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A (Experimental): Avelumab plus External Beam Radiation Therapy (EBRT)
  Interventions: Drug: Avelumab; Radiation: External Beam Radiation Therapy (EBRT)
- Arm B (Experimental): Avelumab plus Lutetium-177 (177Lu)-DOTATATE This treatment arm is now closed to recruitment
  Interventions: Drug: Avelumab; Radiation: Lutetium-177 (177Lu)-DOTATATE

INTERVENTIONS:
Drug: Avelumab — All patients will receive avelumab intravenously (IV) at 10 mg/kg every 2 weeks for 24 months or until unacceptable toxicity or evidence of disease progression
  Other Names: Bavencio; Anti-PD-L1
Radiation: External Beam Radiation Therapy (EBRT) — Patients allocated to Arm A will receive EBRT on 2 occasions, 8-10 weeks apart
  Other Names: Radiotherapy
  Arms: Arm A
Radiation: Lutetium-177 (177Lu)-DOTATATE — Patients allocated to Arm B will receive 177-Lu-DOTATATE treatment on 2 occasions, 8-10 weeks apart.
  This treatment arm is now closed to recruitment.
  Other Names: Peptide Receptor Radionuclide Therapy (PRRT); Lutathera
  Arms: Arm B

SUMMARY:
10.17 GoTHAM is intended as a signal-seeking, biomarker, phase Ib/II study that will evaluate the safety and anti-tumour activities of the novel combination of avelumab with 177-Lu-DOTATATE (a type of peptide receptor radionuclide therapy; PRRT) or external beam radiation therapy (EBRT) in patients with metastatic Merkel cell carcinoma (mMCC).

DETAILED DESCRIPTION:
Despite recent advances with immune checkpoint inhibitors, such as avelumab which has changed the treatment landscape for metastatic Merkel Cell Carcinoma (mMCC), many mMCC patients who attained an initial response exhibit acquired resistance within 1 year. Therefore, novel treatment combinations are needed to improve patient outcome. MCC is an exquisitely radiosensitive tumour and there is emerging data supporting the role of radiation in inducing immunogenic cell death and therefore potentially improving the anti-tumour efficacy when combined with immune checkpoint inhibitors. Peptide receptor radionuclide therapy (PRRT) is used in first-line treatment for neuroendocrine tumours (NETs), by delivering radiation to somatostatin receptor (SSTR) expressing tumour cells. Most NETs, including MCC, express SSTR. Therefore, MCC tumours are ideal candidates for PRRT, and immune checkpoint inhibitor combination approaches with PRRT are highly attractive.

The GoTHAM trial is intended as a signal-seeking and biomarker study. It is designed as a prospective, open-labelled, multi-institutional, two-arm, phase Ib/II trial that will evaluate the safety and anti-tumour activity of 177Lu-DOTA-octreotate (LuTate) or external beam radiation therapy (EBRT) in combination with avelumab in patients with mMCC. The primary objective is to evaluate the anti-tumour activity as reflected by PFS rate at 12 months.

The LuTate arm of this study is now closed to recruitment.

ELIGIBILITY:
Inclusion Criteria:

* Patient is 18 years of age or older and who has provided written informed consent.
* Patient has histologically confirmed metastatic MCC.
* Eastern Cooperative Oncology Group (ECOG) performance status of ≤2 .
* Willing and able to comply with all study protocol requirements for the duration of the study.
* Patient must have measurable disease by CT or MRI per RECIST version 1.1 criteria.
* Patient is treatment naïve (no prior systemic therapy for unresectable or metastatic MCC). Note that prior chemotherapy is permitted in the adjuvant setting for loco-regional disease. Prior radiation is permitted for treatment of the primary or loco-regional disease.
* At least 2 weeks since the completion of prior therapy, including surgery or radiotherapy.
* Screening laboratory values, obtained within 14 days prior to registration/randomisation must meet the criteria specified in the protocol.
* Women of childbearing potential (WOCBP) must use appropriate method(s) of contraception
* WOCBP must have a negative serum or urine pregnancy test within within 7 days prior to the start of avelumab treatment and should be performed every 4 weeks in line with other safety bloods or clinical reviews.
* Male patients who are sexually active with a WOCBP must use any contraceptive method with a failure rate of less than 1% per year.
* Patient must be agreeable to have archival tumour material collected

Exclusion Criteria:

* Patient is excluded if they have ever had any brain or leptomeningeal metastases.
* Prior exposure to immune checkpoint inhibitors (e.g. anti-CTLA-4, anti-PD-1/PD-L1/PD-L2, etc.) or any other antibody or drug specifically targeting T-cell co-stimulation or immune checkpoint pathways.
* Prior exposure to 177Lu-DOTATATE.
* Prior malignancy within the previous 2 years, except for locally curable cancers that have been apparently cured (e.g. basal or squamous cell skin cancer, superficial bladder cancer or carcinoma in situ of the cervix, colon, bladder or breast).
* Life expectancy of 6 months or less.
* An active, known or suspected autoimmune disease that might lead to clinically significant deterioration as per the investigator when receiving an immunostimulatory agent. Patients are permitted to enrol if they have vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger. They are permitted to enrol if they have clinically quiescent auto-immune conditions not requiring immunomodulation beyond low dose steroids (ie <10mg per day of prednisolone or equivalent) or topical therapies (including mesalazine or steroid enemas).
* Current use of immunosuppressive medication, with exceptions detailed in the protocol
* Prior organ transplantation, including allogeneic stem-cell transplantation.
* Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS).
* Positive test for hepatitis B virus (HBV) surface antigen and/or confirmatory hepatitis C virus (HCV) RNA (if anti-HCV antibody tested positive at Screening).
* Pregnant or breastfeeding.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Patients should be excluded if they have a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration.
* Persisting toxicity related to prior therapy (NCI CTCAE v5.0 Grade > 1); however, alopecia, sensory neuropathy Grade ≤ 2, or other Grade ≤ 2 not constituting a safety risk based on Investigator's judgement are acceptable.
* Known prior severe hypersensitivity to investigational product or any component in its formulations, including known hypersensitivity reactions to monoclonal antibodies (NCI CTCAE v5.0 Grade 3).
* Patients with symptomatic or impending cord compression unless appropriately treated beforehand and clinically stable.
* Use of any live vaccines against infectious diseases (e.g., influenza, varicella, etc.) within 30 days of registration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Estimated)
Dates: Start 2020-10-08 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) at 12 months | 3 years
  To evaluate the anti-tumour activity as reflected by PFS rate at 12 months. PFS is defined as the time from treatment initiation until the first date of documented radiographic progression or death due to any cause, whichever occurs first. The radiographic progression will be assessed by the Investigator according to RECIST v1.1.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) at 24 months | 4 years
  Time to disease progression including rate at specific landmark timepoint of 24 months.
Overall Survival (OS) at 12 and 24 months | 4 years
  OS rates at specific landmark timepoints of 12 and 24 months. OS is defined as the time from treatment initiation to the date of death due to any cause.
Best Objective Response Rate (ORR) according to RECIST v1.1 | 4 years
  To evaluate best ORR according to response evaluation criteria in solid tumours version 1.1 (RECIST v1.1). ORR is defined as PR or CR at any stage from time of treatment initiation according to RECIST v1.1.
The safety and tolerability of 177Lu-DOTATATE or EBRT in combination with avelumab. | 4 years
  Rate of treatment-related adverse events (AEs). Safety will be measured by serious adverse events (SAEs) and AEs assessed using the NCI CTCAE v5.0.
Rate of treatment discontinuation due to toxicity | 4 years
  This is defined as the proportion of patients who discontinue with treatment due to treatment-related toxicity.

CONTACTS AND LOCATIONS:
Overall Officials: Prof Shahneen Sandhu, MBBS, FRACP, Study Chair — Peter MacCallum Cancer Centre, Australia
Locations (10):
- Australia (10):
  - Mid North Coast Cancer Institute - Coffs Harbour Health Campus, Coffs Harbour, New South Wales
  - Lake Macquarie Private Hospital, Gateshead, New South Wales
  - Gosford Hospital, Gosford, New South Wales
  - Wyong Hospital, Hamlyn Terrace, New South Wales
  - Royal North Shore Hospital, Sydney, New South Wales
  - Royal Brisbane and Women's Hospital, Brisbane, Queensland
  - Princess Alexandra Hospital, Brisbane, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - Sir Charles Gaidner Hospital, Perth, Western Australia

IPD SHARING:
Plan to Share IPD: No